CLINICAL TRIAL: NCT02245360
Title: A Randomized, Double-blind, Placebo-controlled Study Investigating the Immunologic Effects and Safety of 60-day Treatment of the SQ Grass SLIT-tablet in Adult Subjects With Grass Pollen-induced Allergic Rhinoconjunctivitis
Brief Title: Study Immunology and Safety of 60-day Treatment of SQ Grass SLIT (Sublingual Immunotherapy)-Tablet in Adult Subjects With Grass Pollen-induced Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GRAS3001
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: GRAZAX
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Grazax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grass tablet 75,000 SQ-T (Experimental): Grass tablet 75,000 Standardized Quality units Tablet (SQ-T)
  Interventions: Drug: Phleum pratense grass pollen allergen extract
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Phleum pratense grass pollen allergen extract — Allergy Immunotherapy grass tablet 75,000 SQ-T given once daily over 60 days
  Other Names: GRAZAX/GRASTEK
  Arms: Grass tablet 75,000 SQ-T
Drug: placebo — placebo tablet given once daily over 60 days
  Arms: Placebo

SUMMARY:
To investigate the immunologic effects and safety of 60-day treatment of the Standardized Quality units (SQ) grass Sublingual immunotherapy (SLIT)-tablet in adult subjects with grass pollen-induced allergic rhinoconjunctivitis in a double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* clinical history consistent with grass pollen-induced allergic rhinoconjunctivitis.
* Use of symptomatic treatment of grass pollen-induced allergic rhinoconjunctivitis.
* Positive skin prick test response (wheal diameter ≥3 mm) to Phleum pratense.
* If asthma, daily use of Inhaled corticosteroid (ICS) should be ≤400 microgram budesonide or equivalent
* Moderate or higher level of Phleum pratense specific IgE (Immunoglobulin E) (defined as ≥IgE Class 2; or ≥0.70 Kilo Units/liter (kU/L))

Exclusion Criteria:

* Reduced lung function (defined as FEV1 < 70% (FEV1=Forced Expiratory Volume in 1 second) of predicted value after adequate pharmacologic treatment) measured at Visit 1 and Visit 2
* Clinical history of uncontrolled asthma within 3 months prior to the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Kazei, MD PhD, Study Director — Abbott
Locations (15):
- Russia (15):
  - Research facility ID ORG-001086, Moscow
  - Research facility ID ORG-001018, Moscow
  - Research facility ID ORG-001005, Moscow
  - Research facility ID ORG-001009, Moscow
  - Research facility ID ORG-001016, Moscow
  - Research facility ID ORG-001006, Moscow
  - Research facility ID ORG-001085, Moscow
  - Research facility ID ORG-001014, Moscow
  - Research facility ID ORG-001007, Saint Petersburg
  - Research facility ID ORG-001019, Saint Petersburg
  - Research facility ID ORG-001008, Saint Petersburg
  - Research facility ID ORG-001015, Samara
  - Research facility ID ORG-001021, Saratov
  - Research facility ID ORG-001017, Smolensk
  - Research facility ID ORG-001020, Ufa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Grass Tablet 75,000 SQ-T | Placebo
Started | 53 | 54
Completed | 48 | 52
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grass Tablet 75,000 SQ-T | Placebo | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (11.2) | 34.1 (10.1) | 34.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 26 | 33 | 59
Region of Enrollment [Number; unit: participants]
  Russian Federation | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is Change From Baseline to End of Treatment of Phleum Pratense Specific Immunoglobulin G4 (IgG4) in Serum
Description: measurement of IgG4 in serum
Time Frame: baseline versus end of treatment (approx. 60 days)
Population: In each treatment arm/group 1 subject was excluded from the analyzed sample due to missing post-baseline efficacy data.
Measure: Mean (Standard Deviation); unit: mgA/L
Arm/Group | Grass Tablet 75,000 SQ-T | Placebo
Number analyzed (Participants) | 52 | 53
mgA/L | 0.684 (1.691) | 0.050 (0.588)

2. Secondary Outcome: Change of Phleum Pratense Specific Immunoglobulin E (IgE) From Baseline to End of Treatment
Description: measurement of IgE in serum
Time Frame: baseline versus end of treatment (approx. 60 days)
Population: In each treatment arm/group 1 subject was excluded from the analyzed sample due to missing post-baseline efficacy data.
Measure: Mean (Standard Deviation); unit: UA/ml
Arm/Group | Grass Tablet 75,000 SQ-T | Placebo
Number analyzed (Participants) | 52 | 53
UA/ml | 22.751 (29.364) | -2.756 (16.933)

ADVERSE EVENTS:
Arm/Group | Grass Tablet 75,000 SQ-T | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 26/53 | 12/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grass Tablet 75,000 SQ-T (N=53) | Placebo (N=54)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 4 (4)
Oral pruritus (Gastrointestinal disorders) | 7 (7) | 2 (2)
Tongue oedema (Gastrointestinal disorders) | 3 (3) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 6 (6)
Ear pruritus (Ear and labyrinth disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No